CLINICAL TRIAL: NCT07133113
Title: Medium-term Effects of Treatments in Autoimmune Encephalitis (META): a Real-life, Observational Prospective Study
Brief Title: Medium-term Effects of Treatments in Autoimmune Encephalitis
Acronym: META
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5346
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-03

CONDITIONS: NMDAR Autoimmune Encephalitis; LGI1 Antibody Associated Encephalitis; CASPR2-Antibody; IgLON5; GAD65; GFAP
Keywords: Paraneoplastic neurological disorder; autoimmune encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, DNA, CSF, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- group 1 : Patients with NMDAR encephalitis: Patients with untreated anti-NMDAR encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).
- group 2 : Patients with GAD encephalitis: Patients with untreated anti-GAD encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).
- group 3 : Patients with LGI1 encephalitis: Patients with untreated anti-LGI1 encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).
- group 4 : Patients with IgLON5 encephalitis: Patients with untreated anti-IgLON5 encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).
- group 5 : Patients with GFAP encephalitis: Patients with untreated anti-GFAP encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).
- group 6 : Patients with CASPR2 encephalitis: Patients with untreated anti-CASPR2 encephalitis or with a decision to treat within the previous 30 days
  Interventions: Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression).

INTERVENTIONS:
Other: We aim to assess the clinical response to the treatment initiation protocols most commonly used in autoimmune encephalitis (first-line, first-line with rituximab, dual immunosuppression). — The patients will be identified via the French Nationwide Multidisciplinary Team Meetings for Autoimmune encephalitis, which are conducted on a bi-monthly basis. All patients with newly diagnosed NMDAR, LGI1, CASPR2, IgLON5, GFAP or GAD65 encephalitis and treated for less than 8 weeks will be included. Treatment protocols at the initiation of therapy will be stratified into: 1) first-line only; 2) rituximab without cyclophosphamide; 3) rituximab combined with cyclophosphamide; 4) others.
  The referral clinicians will be contacted by email and the data will be collected using standardized questionnaires, which will be sent at baseline (visit 1, V1) and 4 months after the initiation of therapy (visit 2, V2). The questionnaires will be structured into 7 sections:
  * 1 Demographics
  * 2 Symptoms
  * 3 Cognitive screening tests (MMSE, MoCA, and/or others)
  * 4 Level of dependence (ADL, I-ADL, mRS, CASE) and impact on social life
  * 5 Diagnostic tests (brain MRI, brain PET, CSF, and EEG findings)

SUMMARY:
Autoimmune encephalitides are severe neurological disorders requiring urgent treatment, even though there is no standard guideline by lack of empirical evidence. Commonly used treatments are divided into so-called first-line (steroids, intravenous immunoglobulins, plasma exchanges) and second-line (rituximab, cyclophosphamide, tocilizumab, others), and may be used in association or sequentially. There is no standard practice, and initial treatment protocol may consist in first-line alone, first-line with rituximab, or first-line with dual immunosuppression (rituximab and cyclophosphamide). Absence of clear response to initial treatment in the first 4 to 6 weeks may indicate undertreatment and is generally followed by treatment escalation, mostly to dual immunosuppression. However, as the frequency of non-responders to initial treatment is unknown, it is still unclear whether dual immunosuppression should be offered to all patients from inception.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child patient with encephalitis defined as anti-GAD, NMDAR, LGI1, CASPR2, IgLON5 or GFAP
* Untreated or with a decision to treat within the previous 30 days.

Exclusion Criteria:

- Refusal by the referring doctor to participate or refusal by the patient mentioned in the objection to the use of his/her clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients with autoimmune encephalitis defined anti-GAD NMDAR, LGI1, CASPR2, IgLON5 or GFAP and untreated within the previous 30 days
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Failure of the initial treatment protocol | At baseline and 4 months after the initiation of therapy
  Failure of the initial treatment protocol, reflected by the decision to escalate treatment between V1 and V2. Treatment escalation is defined as the addition of one or more second-line treatments more than 30 days after the start of the initial treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civil de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No